CLINICAL TRIAL: NCT05433870
Title: Inflammatory Biomarkers for the Diagnosis of Obstetric Posterior Reversible Encephalopathy Syndrome
Brief Title: Inflammatory Biomarkers for the Diagnosis of oPRES
Status: Completed | Type: Observational
Sponsor: Dunjin Chen (Other)
Responsible Party: Sponsor-Investigator, Dunjin Chen, Director of obstetrics, Guangzhou Medical University
Organization: Guangzhou Medical University (Other)
Other Study IDs: 2019B08
Record Dates: First submitted 2022-06-16; First posted 2022-06-27 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-06

CONDITIONS: Posterior Reversible Encephalopathy Syndrome; Inflammatory Biomarkers; Neutrophil-lymphocyte Ratio
MeSH Terms: conditions — Posterior Leukoencephalopathy Syndrome | interventions — Pressure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PRES group: patients in PE or E with PRES
  Interventions: Other: Whether the PE or E patient combined with PRES
- NON-PRES group: patients in PE or E without PRES

INTERVENTIONS:
Other: Whether the PE or E patient combined with PRES — According to the Diagnostic criteria of PRES, all the patients grouped into two groups.
  Groups: PRES group

SUMMARY:
The purpose of this study is to explore the inflammatory biomarkers for the diagnosis of obstetric posterior reversible encephalopathy syndrome.

DETAILED DESCRIPTION:
The investigators retrospectively collected data (General information, clinical data, biochemical indicators, imaging features, and pregnancy outcome) from pregnant woman diagnosed with PRES to explore the inflammatory biomarkers for the diagnosis of oPRES during 2012 to 2021.Then, the investigators grouped all the patients into PRES group (PE or E with PRES) and NOT-PRES group (PE or E without PRES) according to the diagnostic criteria of PRES. Then, the investigators analysed the inflammatory biomarkers, such as neutrophil-lymphocyte ratio (NLR), platelet-lymphocyte ratio (PLR), monocyte-lymphocyte ratio (MLR), and so on of two groups, and compared the difference of tow groups.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women were diagnosed of PE or E.
2. All patients were examined the cranial imaging (MRI or CT), and imaging findings meeting the diagnostic criteria of PRES or normal.
3. all patients provided written informed consent.

Exclusion Criteria:

1. patients combined with other neurological disorders
2. patients combined with mental illness

Ages: 16 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pregnant Women diagnosed with PE or E.
Sampling Method: Non-Probability Sample
Enrollment: 621 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
inflammatory biomarkers | Inflammatory biomarkers were collected within 1 day after the onset of symptoms.
  The values of neutrophil-lymphocyte ratio, platelet-lymphocyte ratio and monocyte-lymphocyte ratio will be measured.
cranial Imaging | Cranial Imaging was examined within 3 days after the onset of symptoms, such as s headaches, visual changes, seizures, consciousness impairment.
  According to the cranial Imaging, PE or E patients were grouped into PRES group (typical features presence of vasogenic edema in the white matter of the portions of both cerebral hemispheres) and NOT-PRES group (imaging findings were normal).

SECONDARY OUTCOMES:
other biochemical parameters | biochemical parameters were collected within 1 week of the hospital stay.
  The levels of C-Reactive protein (CRP) will be measured,and CRP﹥8000μg/L means a worse outcome.
Blood Pressure(BP) | The BP of patients was obtained within 1hour after the onset of symptoms.
  blood pressure including systolic blood pressure (SBP), and diastolic blood pressure (DBP).
pregnancy outcomes | The pregnancy outcomes will record immediately when the patients deliver.
  The rates of stillbirth and premature birth (gestation less than 37 weeks) in PRES patients.

CONTACTS AND LOCATIONS:
Overall Officials: Dunjin Chen, Principal Investigator — The Third Affiliated Hospital of Guangzhou Medical University
Locations (1):
- Department of Obstetrics and Gynecology, Key Laboratory for Major Obstetric Diseases of Guangdong Province, The Third Affiliated Hospital of Guangzhou Medical University, Guangzhou, China

IPD SHARING:
Plan to Share IPD: No